CLINICAL TRIAL: NCT07098364
Title: A Phase 1/2 Open-Label Study Evaluating the Safety and Efficacy of ST-067 in Combination With CD19-Directed CAR T-Cell Therapy in Patients With Relapsed/Refractory (R/R) Large B-Cell Lymphoma (LBCL)
Brief Title: ST-067 in Combination With CD19-Directed CAR T-Cell Therapy (Liso-cel) in Relapsed/Refractory Large B-Cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Simcha Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1125654; NCI-2025-04890 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20817 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Recurrent Grade 3b Follicular Lymphoma; Recurrent High-Grade B-Cell Lymphoma; Recurrent Indolent B-Cell Non-Hodgkin Lymphoma; Recurrent Primary Mediastinal Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Refractory Grade 3b Follicular Lymphoma; Refractory High-Grade B-Cell Lymphoma; Refractory Indolent B-Cell Non-Hodgkin Lymphoma; Refractory Primary Mediastinal Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Biopsy; Leukapheresis; Spinal Puncture; Magnetic Resonance Spectroscopy; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (liso-cel, ST-067) (Experimental): Patients undergo leukapheresis and lymphodepleting chemotherapy between days -5 to -3 prior to treatment and receive liso-cel IV on day 0. Patients then receive ST-067 SC weekly on days 14, 21, and 28 or days 10, 17, and 24. Patients may continue to receive maintenance ST-067 SC at day 35 once weekly. Treatment continues for up to 8 doses in the absence of disease progression or unacceptable toxicity. Patients undergo x-ray imaging, and ECHO or MUGA during screening. Patients also undergo CT and/or PET as well as lumbar puncture for CSF collection and bone marrow aspiration and biopsy as clinically indicated during screening and follow-up. Patients undergo blood sample collection throughout the study.
  Interventions: Biological: Vevoctadekin; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Leukapheresis; Biological: Lisocabtagene Maraleucel; Procedure: Lumbar Puncture; Procedure: Lymphodepletion Therapy; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Procedure: X-Ray Imaging; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: Vevoctadekin — Given SC
  Other Names: ST-067; ST 067; ST067; Variant ST-067; Engineered IL-18 Variant ST-067; Engineered Interleukin-18 Variant ST-067
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocyte Adsorptive Apheresis; Leukocytopheresis; Therapeutic Leukopheresis; White Blood Cell Reduction Apheresis
Biological: Lisocabtagene Maraleucel — Given IV
  Other Names: Anti-CD19-CAR Genetically Engineered Autologous T Lymphocytes JCAR017; Anti-CD19-CAR Genetically Engineered Autologous T-lymphocytes JCAR017; Autologous Anti-CD19-EGFRt-4-1BB-zeta-modified CAR CD8+ and CD4+ T-lymphocytes JCAR017; Breyanzi; JCAR 017; JCAR-017; JCAR017; Liso-cel
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Lymphodepletion Therapy — Undergo lymphodepletion chemotherapy
  Other Names: Lymphodepleting Therapy; Lymphodepletion
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: X-Ray Imaging — Undergo x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray
Procedure: Biospecimen Collection — Undergo blood and CSF sample collection
  Other Names: Biological Sample Collection

SUMMARY:
This phase I/II trial tests the safety, side effects, and best dose/regimen of ST-067 in combination with CD19-directed chimeric antigen receptor (CAR) T-cell therapy (liso-cel) and how well it works in treating patients with large B-cell lymphoma (LBCL) that has come back after a period of improvement (recurrent) or LBCL that has not responded to previous treatment (refractory). ST-067 is an engineered variant of the human cytokine interleukin-18 that may help the immune system kill cancer cells. Lisocabtagene maraleucel (liso-cel) is an autologous CAR T-cell therapy prepared using the person's own immune system (a group of cells, tissues, and organs that protect the body from attack by bacteria, viruses, and cancer cells) to fight the cancer. Giving ST-067 in combination with liso-cel may better treat patients with relapsed/refractory LBCL.

DETAILED DESCRIPTION:
OUTLINE: This is a phase I, dose-escalation study of ST-067 followed by a phase II study.

Patients undergo leukapheresis and lymphodepleting chemotherapy between days -5 to -3 prior to treatment and receive liso-cel intravenously (IV) on day 0. Patients then receive ST-067 subcutaneously (SC) weekly on days 14, 21, and 28 or days 10, 17, and 24. Patients may continue to receive maintenance ST-067 SC at day 35 once weekly. Treatment continues for up to 8 doses in the absence of disease progression or unacceptable toxicity. Patients undergo x-ray imaging, and echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening. Patients also undergo computed tomography (CT) and/or positron emission tomography (PET) as well as lumbar puncture for cerebral spinal fluid (CSF) collection and bone marrow aspiration and biopsy as clinically indicated during screening and follow-up. Patients undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 3, 6, 9, and 12 months after CAR T-cell infusion, then will be followed per standard of care long-term follow-up until the patient dies, is lost to follow-up, or withdraws consent.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >= 18 years of age at the time of consent
* Patients with LBCL (including diffuse large B-cell lymphoma [DLBCL] not otherwise specified [including DLBCL arising from indolent lymphoma], high-grade B-cell lymphoma, primary mediastinal large B-cell lymphoma, and follicular lymphoma grade 3B) with at least 2 lines of systemic therapy and an Food and Drug Administration (FDA)-approved indication for treatment with liso-cel
* Fluorodeoxyglucose (FDG)-avid disease on PET imaging before lymphodepletion or pathology evidence of active disease
* Evidence of CD19 expression on any prior or current tumor specimen or a high likelihood of CD19 expression based on disease histology
* Karnofsky performance status >= 60%
* Adequate bone marrow function for lymphodepletion chemotherapy defined as: absolute neutrophil count (ANC) >= 1000 cells/mm^3, platelets >= 50,000 cells/mm^3, and hemoglobin >= 8 g/dL, unless the cytopenias are due to bone marrow involvement by lymphoma in the opinion of the principal investigator (PI)
* Calculated creatinine clearance (Cockcroft/Gault) > 30 mL/min/1.73 m^2
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN) (or < 5 x ULN for subjects with lymphomatous infiltration of the liver) and total bilirubin =< 2 (or < 3.0 for subjects with Gilbert's syndrome, lymphomatous infiltration of the liver, or hemolysis)
* Adequate pulmonary function based on pulmonary function testing (PFT), defined as forced expiratory volume in 1 second (FEV1) and FEV1/forced vital capacity (FVC) ratio of >= 60% of predicted value and diffusing capacity of the lung for carbon monoxide (DLCO; corrected) >= 40% of predicted value
* Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) >= 40% as assessed by echocardiogram or multiple uptake gated acquisition (MUGA)
* Women of reproductive potential (defined as all women physiologically capable of becoming pregnant) must agree to use suitable methods of contraception for at least 30 days after the last dose of study therapy (ST-067)
* Males who have partners of reproductive potential must agree to use an effective barrier contraceptive method for at least 90 days after the last dose of study therapy (ST-067)
* Ability to understand and provide informed consent
* Able and willing to comply with study visit schedule and procedures, including tumor biopsy where feasible and with acceptable risk

Exclusion Criteria:

* Planned use of out-of-specification liso-cel product
* History of another malignancy. The following are exceptions to this criterion:

  * Adequately treated basal cell or squamous cell carcinoma of the skin.
  * In situ prostate, ductal breast carcinoma breast, and cervical carcinoma.
  * Adequately treated papillary, noninvasive bladder cancer.
  * Other adequately treated stage 1 or 2 cancers currently in complete remission.
  * Any other cancer that has been in remission for >= 2 years
* Planned use of therapeutic doses of corticosteroids (> 20 mg/day prednisone or equivalent) or other systemic immunosuppression within 7 days prior to leukapheresis or within 72 hours prior to liso-cel infusion. Topical and/or inhaled steroids are permitted
* Prior treatment with any CD19 CAR T-cell therapy
* For allogeneic hematopoietic cell transplant recipients, active graft versus host disease (GVHD) and/or systemic GVHD therapy within 30 days prior to planned leukapheresis
* Known active hepatitis B (detectable hepatitis B deoxyribonucleic acid [DNA]) or hepatitis C (detectable hepatitis C ribonucleic acid [RNA])
* Known human immunodeficiency virus (HIV) infection
* Pregnant or breastfeeding women
* Prior treatment with any IL-1 or IL-18 agonist and/or biosimilar agents, or an investigational agent within 4 weeks or 5 half-lives, whichever is shorter, prior to start of lymphodepletion
* Active autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., ulcerative colitis, Crohn's disease], celiac disease, or other serious chronic gastrointestinal conditions associated with diarrhea, autoimmune vasculitis, systemic lupus erythematosus, Wegener syndrome [granulomatosis with polyangiitis], myasthenia gravis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.) requiring immunosuppressive therapy. The following are exceptions to this criterion:

  * Vitiligo.
  * Alopecia.
  * Hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.
  * Type 1 diabetes mellitus.
  * Psoriasis not requiring systemic treatment.
  * Conditions considered to be low risk of serious deterioration by the PI
* History of any one of the following cardiovascular conditions within the past 6 months, unless clearance by a cardiologist is obtained: class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, or unstable angina. History of other clinically significant cardiac disease that, in the opinion of the PI or designee, is a contraindication to study treatment is also excluded
* Significant electrocardiogram (ECG) abnormalities, including unstable cardiac arrhythmia requiring medication, second-degree atrioventricular (AV) block type II, third-degree AV block, >= grade 2 bradycardia, or QT interval corrected using Fridericia's formula > 500 ms irrespective of gender
* History or presence of clinically relevant central nervous system (CNS) pathology, such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, or psychosis that in the opinion of the PI is a contraindication to study treatment.

  * Patients with active parenchymal CNS involvement by malignancy will be excluded. Patients with prior or current secondary leptomeningeal CNS disease are eligible. CNS disease prophylaxis must be stopped at least 1 week prior to liso-cel infusion
* History of solid organ transplantation
* Active, serious, and uncontrolled infection(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-12-27 (Actual); Primary Completion 2030-10-04 (Estimated); Study Completion 2043-10-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 4 years
  Will be graded in severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, with the exception of cytokine release syndrome and immune effector cell-associated neurotoxicity syndrome, which will be graded according to the American Society for Transplantation and Cellular Therapy consensus criteria. The type, frequency, and severity of AEs and laboratory abnormalities will be listed and summarized.
Dose limiting toxicities (DLT) | Up to 21 days following the first vevoctadekin (ST-067) dose
  Will be graded in severity according to the NCI CTCAE version 5.0. Will be summarized based on the DLT evaluable population. Final DLT rates at each dose level will be estimated by isotonic regression by applying the pooled adjacent violators algorithm. The target toxicity rate is 30%.
Optimal biological regimen | Up to 4 years
  Will be assessed based on safety and tolerability, confirmation of maximum target engagement, optimal biological effects without undesirable clinical effects, pharmacokinetics parameters, and biological response data.
Complete response (CR) rate | At 3 months after liso-cel infusion
  Will be assessed by Lugano criteria. Will be summarized along with the 2-sided 95% exact Clopper-Pearson confidence interval (CI) based on the efficacy-evaluable population.

SECONDARY OUTCOMES:
CR rates | At 6 months after liso-cel infusion
  Will be assessed by Lugano criteria. Will be summarized along with the 2-sided 95% exact Clopper-Pearson CI based on the efficacy evaluable population.
Overall response rates | At 6 months after liso-cel infusion
  Will be assessed by Lugano criteria. Will be summarized along with the 2-sided 95% exact Clopper-Pearson CI based on the efficacy evaluable population.
Duration of response (DOR) | Up to 4 years
  DOR will be assessed among responders. If a patient does not have an event for the DOR analyses, the patient will be censored at the date of the last adequate disease assessments or prior to the earliest censoring event. The censoring reason can include last contact/follow-up, discontinuation or completion of the study, receipt of another anticancer treatment with the exception of consolidation therapy with hematopoietic cell transplantation (HCT), and at least two consecutive missed scheduled disease assessments. Kaplan-Meier (KM) method will be used.
Progression free survival (PFS) | Up to 4 years
  If a patient does not have an event for the PFS analyses, the patient will be censored at the date of the last adequate disease assessments or prior to the earliest censoring event. The censoring reason can include last contact/follow-up, discontinuation or completion of the study, receipt of another anticancer treatment with the exception of consolidation therapy with HCT, and at least two consecutive missed scheduled disease assessments. KM method will be used.
Overall survival (OS) | Up to 4 years
  Analyses of OS will be performed in the safety population. For assessment of OS, data from surviving patients will be censored at the last time that the patient is known to be alive. KM method will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre V. Hirayama, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No